CLINICAL TRIAL: NCT06645574
Title: Towards a Health Promotion for Children Engaged in Sport Intensive Practice for a Healthy Adult
Acronym: PROTEGE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondation Lenval (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 24-HPNCL-04
Record Dates: First submitted 2024-10-15; First posted 2024-10-17 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Prevention
MeSH Terms: interventions — Physical Therapists

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Girls practizing gymnastics 8 to 15 yo (Experimental)
  Interventions: Other: The multidisciplinary preventive approach among young people involved in intensive sports activities. Athlete will see doctor and physiotherapist.

INTERVENTIONS:
Other: The multidisciplinary preventive approach among young people involved in intensive sports activities. Athlete will see doctor and physiotherapist. — Athletes will have 2 times per years prevention examination:
  * A standard medical examination
  * A physiotherapy assessment with strength assessment
  * They will complete psychometric evaluation self-questionnaires

SUMMARY:
This project aims to elucidate the complexities of the preventive approach among young people involved in intensive sports activities, providing valuable recommendations to optimize their physical, mental, and social health both in the present and in the long term. The multidisciplinary skills of a team of researchers in sports science and health will contribute their recognized disciplinary expertise through international publications, as well as solid experience in the demands of elite sports, along with a commitment to transferring innovative knowledge toward a preventive approach to sports training.

The main objective is to determine whether a somatotype aligned with the discipline's expectations protects the athlete in terms of self-perception and, consequently, reduces health-risk behaviors. Secondary objectives will include linking somatotype, growth, psychological changes (self-perception), and the emergence of health-risk behaviors or injuries in these young athletes.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 8 to 15 years old
* Intensive athletes: that is to say they practice a competitive sporting activity with a number of hours of weekly training greater than their age in years.(For example, a 10 year old child will need to train more than 10 hours per week to be included.)
* Sport at an early age
* Obtaining written and signed informed consent from one of the two parents or the holder of parental authority
* Affiliation to a social security system

Exclusion Criteria: menstruation for more than a year at the time of inclusion

-

Ages: 8 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 90 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2032-12 (Estimated); Study Completion 2032-12 (Estimated)

PRIMARY OUTCOMES:
Determine whether a somatotype in harmony with the expectations of the discipline protects the athlete in terms of self-perceptions and, consequently, reduces risky behaviors for her health. | 2 times a year for up to 84 months of follow-up
  frequency of occurrence of risky behavior depending on the somatotype of the athletes

SECONDARY OUTCOMES:
1. How does the somatotype of athletes change over time and in response to training? Are these modifications uniform among athletes of the same sex practicing the same sport? | 2 times a year for up to 84 months of follow-up
  The evolution of the somatotype of athletes over time and in response to training Relationship between athlete somatotype and growth acceleration at puberty Self-esteem and perception of physical appearance between athletes conforming and nonconforming to the ideal somatotype of their sport The prevalence of ACAD and excessive training practices among athletes with low self-esteem related to their physical appearance.
  Correlation between athletes' somatotype and their predisposition to health problems, such as eating disorders and sports injuries